CLINICAL TRIAL: NCT03600194
Title: Pilot Study Comparing the Effectiveness of Two Different Methods of Acoustic Stimulation to Enhance Slow Wave Sleep
Brief Title: Pilot Study Comparing the Effectiveness of Two Different Methods of Acoustic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AI-16052-PSCOMP-LO
Record Dates: First submitted 2018-06-28; First posted 2018-07-26 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Sleep Deprivation; Insufficient Sleep Syndrome; Healthy
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, sham-controlled pilot cross-over trial comparing
Who Masked: Participant
Masking Description: Participants will wear a PSG both nights, the set-up between devices will not be the same, but similar
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- PowerSleep Stim (Active Comparator): In this arm soft audio tones (below 65dB) will be administered by the PowerSleep Stim Device during deep sleep as determined by the functionality of the device.
  Interventions: Device: PowerSleep Stim
- PowerSleep Sham (Placebo Comparator): This PowerSleep Sham device is the same as the PowerSleep Stim device, however, it can be configured in a mode that does not play audio tones
  Interventions: Device: PowerSleep Sham
- Northwestern Stim (Active Comparator): The NorthWestern Stim device is set up will function similarly to the PowerSleep prototype. Acoustic stimulation provided by headphones with an audible soft volume that do not result in arousals will be used.
  Interventions: Device: Northwestern Stim
- Northwestern Sham (Placebo Comparator): The Northwestern Sham device will be the same as the Northwestern Stim set up, however no audio tones will be played.
  Interventions: Device: NorthWestern Sham

INTERVENTIONS:
Device: PowerSleep Stim — The PowerSleep Stim device is a wearable and non-invasive device, consisting of a headband with 2 electrodes (one forehead and one mastoid) and speakers covered by foam over each ear. The headband is connected via a tether cable to a user interface which houses the EEG amplifier and electronics of the device. The headband is adjusted via Velcro closure. The device also includes a right mastoid electrode EEG will be recorded by the PowerSleep device. Soft audio tones (below 65dB) will be administered via the speakers system during deep sleep as determined by the functionality of the device. The version being used for this study is considered investigational as this is an earlier version which allows the study team will be able to review EEG data recorded by the PowerSleep device in real time.
  Other Names: SmartSleep
  Arms: PowerSleep Stim
Device: Northwestern Stim — The Northwestern Stim Device will function similarly to the PowerSleep device, but stimulation will be provided using a standard PC (computer) setup at the bedside using standard PSG electrodes. EEG will be monitored and slow wave sleep (SWS) identified using a standard PSG channels (international 10-20 system: Fpz, F3, F4, C3, C4, P3, P4, O1, O2) referenced to left mastoid. Electro-oculogram (EOG) will be recorded using 2 electrodes placed lateral to each eye and chin electromyogram (EMG) was recorded using 3 chin electrodes. The full EEG data set will be collected using Brain Vision Recorder software (Brain Products GmBH) and stored for off-line analysis and sleep scoring. A Matlab script (R2014b, MathWorks, Natick, MA) was developed for online detection of slow-waves and to control acoustic stimulation in a phase-locked manner (targeting the up phase of the slow wave). Acoustic stimulation will be provided by headphones with an audible soft volume that do not result in arousals.
  Arms: Northwestern Stim
Device: PowerSleep Sham — The PowerSleep Sham device is a wearable and non-invasive device, consisting of a headband with 2 electrodes (one forehead and one mastoid) and speakers covered by foam over each ear. The headband is connected via a tether cable to a user interface which houses the EEG amplifier and electronics of the device. The headband is adjusted via Velcro closure. The device also includes a right mastoid electrode EEG will be recorded by the PowerSleep device. There are no audio tones played in the Sham condition. The version being used for this study is considered investigational as this is an earlier version which allows the study team will be able to review EEG data recorded by the PowerSleep device in real time.
  Arms: PowerSleep Sham
Device: NorthWestern Sham — The Northwestern Sham device is set up will function similarly to the PowerSleep prototype. EEG will be monitored and SWS identified using a standard PSG channels (international 10-20 system: Fpz, F3, F4, C3, C4, P3, P4, O1, O2) referenced to left mastoid. Electro-oculogram (EOG) will be recorded using 2 electrodes placed lateral to each eye and chin electromyogram (EMG) was recorded using 3 chin electrodes. The full EEG data set will be collected using Brain Vision Recorder software (Brain Products GmBH) and stored for off-line analysis and sleep scoring. A Matlab script (R2014b, MathWorks, Natick, MA) was developed for online detection of slow-waves. Participant will wear headphones but no audio tones played in the Sham condition.
  Arms: Northwestern Sham

SUMMARY:
This study is a randomized, single-blind, sham-controlled pilot cross-over trial comparing the feasibility, and efficacy of 2 nights of in lab use with active versus sham conditions in adults with sleep restricted schedules. The study involves the testing of 2 different prototypes both in the sham and active conditions The expected duration of the study for each participant is up to 5 weeks. It will include adults (21-50 yr. old) who report shortened sleep due to lifestyle. For the purposes of this study, shortened sleep is defined as sleeping at least 5.5 of sleep per night, and sleeping less than or equal to 7 hours of sleep +/- 15 minutes on at least 3/5 work/school nights. Participants also increase their sleep duration by ≥ 1 hour on non-work/school days. In addition, participants report a sleep latency ≤ 30 minutes and wake after sleep onset ≤ 30 minutes. Participants are generally healthy individuals who have not been diagnosed with any sleep-related medical conditions such as obstructive sleep apnea, insomnia, difficulty falling asleep on a nightly basis and deny difficulty staying asleep if awoken during sleep. In addition, participants diagnosed with major organ system diseases or requiring oxygen therapy are excluded from participation. Up to 60 individuals will be consented in order to complete a total of 10 participants using a cross over design. The study involves an initial screening visit followed by 1 week of actigraphy measurement to determine eligibility. Post eligibility, participants will undergo an additional week of actigraphy measurement. Participants will complete 2 overnight visits in the sleep lab per week, with one washout night in between. They will be randomly assigned to sham or active condition during the first of the overnight visits, and the other condition during the second overnight condition. Participants will return to the lab on the same nights the next week and receive the second device in both conditions. Participants will be asked to complete a battery of cognitive tests upon wake up in the lab after each of the overnight visits.

DETAILED DESCRIPTION:
Each subject will undergo a baseline screening period with screening questionnaires, clinical history, and 1 week of actigraphy measurement to determine eligibility for inclusion in the study. Prior to the overnight study they will undergo an additional 1 week of actigraphy measurement. Each subject will have two 3 day/2 night stays, separated by one week. Including outpatient screening and the inpatient study periods, the duration of participation for each subject will be ~5 weeks. We anticipate 6 months to enroll and complete the 12 subjects. Primary data analysis should be completed within one year of starting this study.

Study Procedures:

Participants may be screened over the phone to determine eligibility. A screening script will include a general review of key inclusion and exclusion criteria, and the Stop-Bang Questionnaire to assess risk for undiagnosed obstructive sleep apnea. Participants that meet all eligibility criteria will be asked to come into the research lab for a brief daytime screening visit. Participants who are interested and eligible will be consented. Participants will be provided with information on use of the actigraph and sleep logs at home. Participants will be asked to return their actigraph and sleep logs to the laboratory either in person or via pre-paid FedEx. Participant qualification will be assessed based on sleep logs and the actigraph results. Qualifying participants will wear the actigraph and fill out sleep logs again for the week prior to their first overnight visit.

Visit 1 (Screening) Procedures (up to 2 hours):

Participants will be asked to report to the research office for a daytime visit. A detailed interview will be performed verifying eligibility criteria, as well as a review of work and non-work schedules. After a full explanation of the protocol and after all the participants questions have been answered, they will be asked to sign the consent form. Written documentation of consent will be obtained for all subjects.

Participants will complete the following baseline questions:

Demographics Medical History Questionnaire Collection of Current Medications Epworth Sleepiness Scale (ESS) Insomnia Severity Index Questionnaire (ISI) (if not completed during telephone screen) Stop-Bang (if not completed during telephone screen) Cambridge Hopkins (Restless Leg Syndrome) Questionnaire (if not completed during phone screen)

Participants will have their height, weight, neck circumference, temperature, heart rate and blood pressure recorded. Women of child bearing potential will have a urine pregnancy test.

Participants will be trained in the use of the sleep logs and actigraphy.

Actigraphy screening:

Participants will be asked to wear an actigraph and complete a daily sleep diary for 7 days +2 days to monitor their sleep schedule. Participants will receive instructions from the study staff on how to wear the actigraph and will be asked to keep to their regular sleep schedule.

Assessment training:

Participants will also be trained on daytime assessments which will be completed during the overnight visits. Only participants that are able to perform the task will be asked to remain in the study and through completion.

Actigraphy review:

Participants will drop off or mail their actigraph and sleep log to the research office for review by the study staff. The actigraph data will be reviewed by a trained technologist. Only participants that demonstrate a regular sleep schedule and an average sleep duration of 6-7 hours during the work week will be asked to return to the lab for the study. A regular sleep schedule will be defined as a bedtime between 9pm and midnight with no more than 1 hour of variability across the 7 nights. Qualifying participants will be asked to continue wearing the actiwatch and completing the sleep diary throughout the remainder of the study.

Visit 2 Procedures (3 days/2 nights with washout in between nights):

Participants will be randomly assigned to the sham or active stimulation condition during the first night of the overnight visits, and the other condition (sham or active stimulation) during the second night of the overnight visits. Participants may also be asked to undergo additional night study testing if data collected is unable to be analyzed due to unforeseen technical or environmental reasons. Participants and study staff will be blinded to the condition they are receiving during each overnight study for prototype 1. However, study staff will not be blinded during each overnight for prototype 2.

Active condition: Participants will be set-up with one of the PowerSleep Prototypes. Soft audio tones (below 65dB to prevent arousals from sleep) will be administered via the headphones during deep sleep throughout the night.

Sham condition: Participants will be set up with the same PowerSleep prototype as with the active arm, however no audio tones will be played.

Participants will typically be asked to arrive at the Sleep Lab ~3 hours before their usual bedtime.

Upon arriving at the sleep lab for the first overnight study, the actigraph data will be downloaded for review by a trained technologist. Only participants that demonstrate a regular sleep schedule and a sleep duration of 6-7 hours per night will be asked to remain in the study and through completion.

The Paired Associated Learning (PAL) learning set will be completed before the participant goes to bed.

Overnight monitoring:

Participants will complete an attended overnight polysomnogram (PSG). During all PSGs, the electroencephalogram (EEG), electrooculogram (EOG) and sub-mental electromyogram (EMG) will be recorded with surface electrodes according to American Academy of Sleep Medicine (AASM) standards. In addition, surface ECG electrodes (standard lead II) will be applied to the participant. All PSG signals will be recorded and monitored continuously by a trained sleep technologist throughout the night.

After the baseline recordings while awake, the PSG channels indicated above will be recorded for the participants' entire night of sleep. Participants will be in a private room with the door closed and lights off. During the overnight recordings, participants will be directly observed via video camera. The participant can contact the trained technologist present at any time via an intercom.

During overnight studies under the active condition, soft auditory tones will be provided via the speakers during N3 sleep for prototype 1 and N2 or N3 sleep for prototype 2.

Morning:

The participant will be awakened at their usual wake time according to sleep logs and actigraphy

Participants will be asked to complete daytime assessments each morning of the visit (90 minutes post awakening) including:

Karolinska Sleepiness Scale (KSS) Samn & Perelli Fatigue Scale Visual Analog Scale (VAS) sleep quality Matrix Reasoning Task (MRT) (to be completed on iPad) Digit Symbol Substitution Task (DSST) (to be completed on iPad) Psychomotor Vigilance Test (PVT-B - 3min) (to be completed on iPad) Paired Associates Learning (PAL)

The DSST, MRT, PVT-B and PAL assessments will be completed electronically and the other assessments will be completed in paper form.

The actigraph data will be downloaded and the re-configured actigraphy device will be returned to the participant to be worn for the period before Visit 4. Sleep logs will be given for the participant to fill out during any time at home.

The subject will be allowed to go home or to work during the day and will be instructed not to nap during the day. This will be monitored with the actigraph. The subject will return to the lab the following evening 3 hours before the usual bedtime and will be instrumented and studied as described for night 1. For example, participants that spent the night Monday and completed Tuesday morning testing will come into the lab Wednesday night for Thursday morning testing or if participants sent Tuesday night and completed Wednesday morning testing they will come into the lab Thursday night for Friday morning testing.

Visit 4 Procedures (3 days/2 nights):

Participants will return to the Sleep Disorders Center to complete the second set of overnight studies one or two weeks after the first set of overnight studies. If participants spent Monday and Wednesday night in the lab for the first set of overnight studies, they will complete the second set of overnight visits Monday and Wednesday. The actigraph data will be similarly downloaded and reviewed for further participation upon arriving at the Sleep Disorders Center. This visit will be identical to Visit 3 except that the subjects will receive the prototype system that was not used in Visit 3 (Prototype 1 or 2).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to admission
* Able to read, write and speak English
* Adult volunteers aged 21-50
* Working full time (M-F) schedule [Note: Full time is considered a 32 hour work week start time at 7am or later] or full time student
* Self-reported regular sleep schedule who are able to maintain their sleep schedule during the course of the study
* Self-reported sleep latency ≤ 30 minutes
* Self-reported wake after sleep onset ≤ 30 minutes
* Participants who regularly (3 of 5 work/school nights) use an alarm clock during the work/school week and who self-report:

  * Regular sleep schedule of 5.5-7 hours +/- 15 minutes on work/school nights [confirmed by actigraphy at visit 2, at least 3 of 5 work/school nights between 5.5 to 7 hours total sleep time]
  * Regular increase in sleep duration by ≥ 1 hour during non-work/school days as compared to work days, either by nocturnal bedtime extension or via a daytime nap [confirmed by actigraphy with at least 1 hour of increased sleep duration during one non-work/school night]
* Participants who demonstrate successful performance of the Paired Associates Learning Task during the training session

Exclusion Criteria:

* Participation in another interventional study in the past 30 days.
* Major controlled* or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, Chronic Obstructive Pulmonary Disease (COPD), respiratory failure or insufficiency, or patients requiring oxygen therapy (as determined by self-report and reviewed by the study PI.)
* History of current or recent (e.g. within past 5 years) narcotic, or any other drug abuse.
* Daily caffeine intake > 650mg
* Current smoker (more than 6 cigarettes a week) or those using nicotine replacement therapy. Those that have been nicotine free for 30 days will be included.
* Currently working night shift, split shift or rotating shift (which includes night shifts).
* Current use, or use within the past month, of a prescription or over-the-counter sleep medication or stimulant; or use of psychoactive medication (based on self-report and review with a study clinician) Refer to table below for examples.
* Individuals who self-report a current severe or chronic medical condition that may affect sleep patterns (based on self-report and review with a study clinician).
* Pregnant or currently breast feeding
* Body Mass Index > 40 kg/m2
* Prior diagnosis (via self report) of any sleep disorder including:

  * Obstructive Sleep Apnea (OSA) (AHI ≥15 events/hour) - from ambulatory or in lab polysomnography
  * Restless legs syndrome, or periodic limb movement disorder
  * Insomnia
  * Parasomnia
  * Circadian Rhythm Sleep-Wake Disorders
* High Risk of OSA based on STOP-BANG Questionnaire ("yes" on at least 4 of 8 questions)
* High risk of Restless Legs syndrome (RLS) base on Cambridge-Hopkins Screening Questionnaire
* High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher)
* Self-reported history of excessive alcohol intake - self-report > 21 drinks/week or binge alcohol consumption (>5 drinks per day)
* Individuals who self-report a history of recurrent seizures or epilepsy or family history of hereditary epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Individuals who self-report severe contact dermatitis or allergy to silicone.
* Individuals who self-report moderate hearing loss.
* Inability to achieve appropriate headband fit (for prototype 1).
* Planned air travel or travel across more than one time zone during the anticipated period of the study with PowerSleep or PLL (Northwestern University) device use.
* Alpha-delta sleep on the first night in the sleep lab.
* Intentional naps during the work week.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No, This data will remain with Northwestern and Philips.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because of all of the different randomization variations, participants could have received the powersleep or the northwestern device first and then could have been randomized to stim or sham first for both set of devices, data has been presented by device rather than overnight device configurations.
Groups:
- All Participants Consented: All participants consented to the study but not enter into the In-lab phase.
- PowerSleep First, Northwestern Second: Participants in this arm received the PowerSleep device first and the Northwestern device second. Participants were randomized to receive PowerSleep Stim or Sham first. Participants and study staff were blinded to assignment. In this arm soft audio tones (below 65dB) will be administered by the PowerSleep Stim Device during deep sleep as determined by the functionality of the device. T
  PowerSleep Stim: The PowerSleep Stim device is a wearable and non-invasive device, consisting of a headband with 2 electrodes (one forehead and one mastoid) and speakers covered by foam over each ear. The headband is connected via a tether cable to a user interface which houses the EEG amplifier and electronics of the device. The headband is adjusted via Velcro closure. The device also includes a right mastoid electrode EEG will be recorded by the PowerSleep device. Soft audio tones (below 65dB) will be administered via the speakers system during deep sleep as determined by the functionality of the device. The version being used for this study is considered investigational as this is an earlier version which allows the study team will be able to review EEG data recorded by the PowerSleep device in real time.
  PowerSleep Sham: the same device as stim with audio turned off.
- Northwestern First, PowerSleep Second: In this arm participants were randomized to received Stim or Sham of the Northwestern device first and the PowerSleep device second. The NorthWestern Stim device is set up will function similarly to the PowerSleep prototype. Acoustic stimulation provided by headphones with an audible soft volume that do not result in arousals will be used.
  Northwestern Stim: The Northwestern Stim Device will function similarly to the PowerSleep device, but stimulation will be provided using a standard PC (computer) setup at the bedside using standard polysomnogram (PSG) electrodes. EEG will be monitored and slow wave sleep (SWS) identified using a standard PSG channels (international 10-20 system: Fpz, F3, F4, C3, C4, P3, P4, O1, O2) referenced to left mastoid. Electro-oculogram (EOG) will be recorded using 2 electrodes placed lateral to each eye and chin electromyogram (EMG) was recorded using 3 chin electrodes. The full EEG data set will be collected using Brain Vision Recorder software (Brain Products GmBH) and stored for off-line analysis and sleep scoring. A Matlab script (R2014b, MathWorks, Natick, MA) was developed for online detection of slow-waves and to control acoustic stimulation in a phase-locked manner (targeting the up phase of the slow wave). Acoustic stimulation will be provided by headphones with an audible soft volume that do not result in arousals.
  Northwestern Sham: Exact same set-up as the stim version but with audio tones turned off.
Period: Screening
Arm/Group | All Participants Consented | PowerSleep First, Northwestern Second | Northwestern First, PowerSleep Second
Started | 38 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 27 | 0 | 0
Period: In Lab Phase
Arm/Group | All Participants Consented | PowerSleep First, Northwestern Second | Northwestern First, PowerSleep Second
Started | 0 | 5 | 6
Completed | 0 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Screening Population: All participants that were consented.
Arm/Group | Screening Population
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 17
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: The Effects of the Auditory Stimulation on the Cumulative or Average Slow-wave Activity (SWA) Delivered by the PowerSleep & Northwestern Systems in Adults With Mildly Sleep Restricted Schedules as Determined by Device and PSG Scoring Outputs.
Description: It is hypothesized that one night of in-lab use of a PowerSleep system (Prototype 1) or NorthWestern (Prototype 2) under an active condition (tones played to increase slow-wave activity), as compared to one night of in-lab use of the same PowerSleep system (prototype 1) or Prototype 2 under a sham condition (no tones played) will result in a significant increase (≥ 5%) in cumulative or average slow-wave activity (SWA) in nonREM sleep across the whole night of sleep compared to sham. Note: The relative ability of Prototype 1 versus Prototype 2 to increase the magnitude of SWA in sleep will also be compared.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: microvolts^2
Arm/Group | PowerSleep Stim | PowerSleep Sham | Northwestern Stim | Northwestern Sham
Number analyzed (Participants) | 11 | 11 | 11 | 11
microvolts^2 | 2083.9 (1229.7) | 1830.9 (975.5) | 2317.0 (1272.2) | 1723.1 (806.3)
Statistical Analysis 1: Comparison: PowerSleep Stim vs PowerSleep Sham vs Northwestern Stim vs Northwestern Sham; Test type: Superiority; p = .019, Mixed Models Analysis; Design*Therapy interaction term

2. Secondary Outcome: The Effects of Active and Sham Conditions of PowerSleep and Northwestern University Systems on Psychomotor Vigilance Task - Brief
Description: The secondary aim of the study is to assess the impact of active versus sham PowerSleep and NorthWestern systems on measures of daytime function (Psychomotor Vigilance Task - Brief ).The Psychomotor Vigilance Task is a sustained-attention, reaction-time task that measures the speed with which participants respond to a visual stimulus. The score is fastest reaction time during a 3 minute assessment.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | PowerSleep Stim | PowerSleep Sham | Northwestern Stim | Northwestern Sham
Number analyzed (Participants) | 11 | 11 | 11 | 11
milliseconds | 310.7 (202.6) | 245.6 (37.0) | 247.4 (43.6) | 248.6 (41.3)

3. Secondary Outcome: The Effects of Active and Sham Conditions of PowerSleep and Northwestern University Systems on Paired Associated Learning
Description: The secondary aim of the study is to assess the impact of active versus sham PowerSleep and NorthWestern systems on measures of daytime function (Paired Associated Learning). The Paired Associates Learning Task is a well-established cognitive task used to assess declarative memory. Participants are presented with word pairs to learn. Immediately following and again in the morning after they wake up they are tested on the recall of the words. The recall testing involves showing participants one word and they are asked to state the paired word that they learned previously. Overnight memory retention is determined by the difference in the number of recalled words between morning retrieval testing after sleep and immediate recall performance at learning before sleep. The testing is scored by a technician and may also be recorded for scoring confirmation. The score is the difference between the post wake up test and evening recall test.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: words
Arm/Group | PowerSleep Stim | PowerSleep Sham | Northwestern Stim | Northwestern Sham
Number analyzed (Participants) | 11 | 11 | 11 | 11
words | 8.7 (7.4) | 10.2 (8.8) | 12.4 (11.7) | 13.1 (9.6)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Screening Population | PowerSleep Stim | PowerSleep Sham | Northwestern Stim | Northwestern Sham
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/38 | 0/11 | 1/11 | 0/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Population (N=38) | PowerSleep Stim (N=11) | PowerSleep Sham (N=11) | Northwestern Stim (N=11) | Northwestern Sham (N=11)
Influenza (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergies (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03600194/Prot_SAP_001.pdf